CLINICAL TRIAL: NCT07166718
Title: Correlation of Pulse Oximetry With Arterial Blood Gas Derived Oxygen Saturation in ICU Patients on Supplemental Oxygen - A Prospective Cross-sectional Study
Brief Title: Running Title: Correlation Between Pulse Oximeter (SpO2) and ABG (SaO2)
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sumit Shahi, Dr, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: BPandey23
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypoxemia; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This was a prospective cross-sectional observational study conducted among 152 patients, admitted to Medical Intensive Care Unit (MICU), who required supplemental oxygen during hospital stay. The ABG analysis was done, and pulse oximeter reading was recorded simultaneously. The goal of the study was to correlate oxygen saturation measured by pulse oximeter (SpO2) with arterial blood gas analysis (SaO2).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in MICU requiring supplemental oxygen

Exclusion Criteria:

* Patients party not giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in MICU of Chitwan medical college, Chitwan requiring supplemental oxygen.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | 3 months
  Correlation between hypoxemia and hypoxia

CONTACTS AND LOCATIONS:
Locations (1):
- Sumit Shahi, Lalitpur, Nepal